CLINICAL TRIAL: NCT03965000
Title: Human SLC5A2 Deficiency and the Glucagon-Incretin Axis: A Pilot Study
Brief Title: Human Solute Carrier Family 5 Member 2 (SLC5A2) Deficiency and the Glucagon-Incretin Axis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 20190121-1930
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Familial Renal Glucosuria; Diabetes Mellitus; Cardiovascular Diseases
Keywords: SGLT2; SLC5A2; glucose metabolism; glucagon; incretin
MeSH Terms: conditions — Glycosuria, Renal; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples acquired during the mixed-meal-tolerance-test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients carrying one or both mutations.
  Interventions: Other: Mixed-meal-tolerance-test
- Controls: Patients not carrying a mutation Familial renal glucosuria causing mutation in the SLC5A2 gene and without impaired glucose tolerance and type 1 or 2 diabetes mellitus.
  Interventions: Other: Mixed-meal-tolerance-test

INTERVENTIONS:
Other: Mixed-meal-tolerance-test — To assess the dynamics of the glucagon-incretin axis we need to perform the MMTT. Thereby the patients need to consume a body weight adjusted, standardized meal and we draw blood at fixed time points over 4 hours.

SUMMARY:
Sodium-glucose-cotransporter 2 (SGLT2) are a new type of oral antidiabetic drugs. SGLT2 inhibitors increase the urinary glucose excretion and thereby decrease blood glucose levels. Beside their glucose lowering effects SGLT2 inhibitors showed beneficial effects on the cardiovascular health. But several studies in cell culture and mice showed that the physiological inhibition of glucagon after meal consumption is impaired when using SGLT2 inhibitors.

The patients carry a rare genetical disease called Familial renal glucosuria (FRG), a human model of life long SGLT2 inhibition. To elucidate the effects of partial and complete SGLT2 inhibition in humans the investigators perform a mixed-meal tolerance test (MMTT), the gold standard for elucidation of insulin and glucagon dynamics.

DETAILED DESCRIPTION:
The index patient was referred to the Department of Internal Medicine I at the Medical University of Innsbruck for evaluation of unclear glucosuria in combination with normal blood glucose levels. The patient suffered from recurrent urinary tract infections and increased urinary frequency, showed a physiological hemoglobin A1c and no further signs of renal dysfunction. Sequencing of the SLC5A2 coding region confirmed that the patient was compound heterozygous for two SLC5A2 mutations. The patient is a mother of five healthy children which are willing to take part in the test. The children show a 50/50 distribution of the mother's mutations. The MMTT will take place after 48 hours of alcohol, sport abstinence and an overnight fasting period. The patients will be given 6 ml/kg body weight of a standardized liquid meal. Blood samples will be collected 10 minutes before consumption of the meal, at the time point of consumption and 15, 30, 60, 120, 150, 180, 210 and 240 minutes after consumption. At each time point six blood tubes will be taken, except at time point -10 and 240 minutes, there is one sample more collected. The investigators aim to assess glucagon, insulin, c-peptide, gastric inhibitory polypeptide (GIP), Glucagon-like peptide-1 (GLP-1), Glucagon-like peptide-2 (GLP-2) levels.

Glucose tolerance will be assessed by using the 4 hours area under the curve (AUC) for glucose. To evaluate the beta-cell function the 4h-AUC's for insulin, c-peptide and the 4h-AUC insulin:glucose ratio will be calculated and compared. The calculation of the alpha-cell function will be performed with the AUC of glucagon and the AUC glucagon/glucose ratio. GIP, GLP-1 and GLP-2 will be determined using the AUC. The AUC's will be calculated by the trapezoidal method.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Capable of giving consent
* One or more SLC5A2 mutations leading to FRG
* Written consent

Exclusion Criteria:

* Impaired glucose tolerance
* Diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One compound heterozygous female index patient and four heterozygous children. The control group consists of age, sex and BMI matched participants from nearly the same area to avoid environmental factors.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the glucagon-incretin axis. | 18 months
  Glucose tolerance will be assessed by using the 4 hours area under the curve (AUC) for glucose.
  Beta-cell function will be assessed by the 4h-AUC's for insulin, c-peptide and the 4h-AUC insulin:glucose ratio will be calculated and compared. The calculation of the alpha-cell function will be performed with the AUC of glucagon and the AUC glucagon/glucose ratio. GIP, GLP-1 and GLP-2 will be determined using the AUC. The AUC's will be calculated by the trapezoidal method
Changes in the gene expression | 18 months
  By collecting blood samples for gene expression analysis before and after the test and comparing it to our healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Rosenstein R, Hough A. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1093-4. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981944
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Bonner C, Kerr-Conte J, Gmyr V, Queniat G, Moerman E, Thevenet J, Beaucamps C, Delalleau N, Popescu I, Malaisse WJ, Sener A, Deprez B, Abderrahmani A, Staels B, Pattou F. Inhibition of the glucose transporter SGLT2 with dapagliflozin in pancreatic alpha cells triggers glucagon secretion. Nat Med. 2015 May;21(5):512-7. doi: 10.1038/nm.3828. Epub 2015 Apr 20. PMID 25894829
- [Background] Pedersen MG, Ahlstedt I, El Hachmane MF, Gopel SO. Dapagliflozin stimulates glucagon secretion at high glucose: experiments and mathematical simulations of human A-cells. Sci Rep. 2016 Aug 18;6:31214. doi: 10.1038/srep31214. PMID 27535321